CLINICAL TRIAL: NCT03640364
Title: Multicenter Prospective Non-randomised Trial of Bilateral Sacrospinous Colposuspension (BSC) in the Treatment of Female Genital Prolapse Accompanied by Urinary Urge Symptomatology
Brief Title: Bilateral Sacrospinous Colposuspension (BSC) in the Female Genital Prolapse With Urinary Urge Symptomatology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helios Medical Center Schleswig (Other)
Responsible Party: Principal Investigator, Dirk G. Kieback, M.D., Ph.D, Head, Dept. of Obstetrics and Gynecology, Helios Medical Center Schleswig
Other Study IDs: HCR051631
Record Dates: First submitted 2018-08-06; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Urinary Urge Incontinence
Keywords: pelvic organ prolapse; incontinence; minimally invasive; vaginal surgery; macroporous; lightweight; mesh; polypropylene; POP; urge
MeSH Terms: conditions — Urinary Incontinence, Urge; Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective non-randomised trial investigating the effect of vaginal vault Suspension on urge symptomatology in female patients with pelvic organ prolapse

DETAILED DESCRIPTION:
A multicenter multinational Trial is performed in 250 female patients with pelvic organ prolapse (POP) and symptoms of urinary urge incontinence.

Dependent on the presence or abscence of the uterus patients are treated with bilateral sacrospinous uterine or vaginal vault suspension (BSC) by means of a tape specifically designed for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* urge urinary incontinence or symptoms thereof
* 18 years old or older
* Compliance regarding data collection, therapy and follow-up
* written informed consent
* simultaneous performance of surgical colporrhaphy permitted

Exclusion Criteria:

* pelvic organ prolapse without symptoms of urinary urge
* age less than 18 years
* no informed consent
* lack of compliance
* adverse reaction to polypropylene
* life expectancy less than anticipated duration of protocol
* ASA 4

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: female patients with pelvic organ prolapse suffering from symptoms of urinary urge incontinence
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Influence of BSC placement on symptoms of urinary urge expressed by change in clinical examination | Checked after 6 weeks, six months and twelve months
  The change in symptoms after the surgical intervention is evaluated by clinical examination . The clinical examination is descriptive, not quantitative and no units are applicable or reportable.
Change in score of standardized ICIQ documentation | Checked after 6 weeks, six months and twelve months
  The International Consultation on Incontinence Questionnaire is used to evaluate Change in Quality of life and urge symptomatology

SECONDARY OUTCOMES:
Anatomical correction of female pelvic organ prolapse | Checked after 6 weeks, six months and twelve months
  Clinical examination of pelvic floor anatomy

CONTACTS AND LOCATIONS:
Overall Officials: Dirk G Kieback, MD,Ph.D, Principal Investigator — Helios Medical Center Schleswig
Locations (1):
- Helios Medical Center, Schleswig, Germany